CLINICAL TRIAL: NCT04984798
Title: Efficacy of Vitamin E in Hyperinsulinism/Hyperammonemia Syndrome
Brief Title: Vitamin E Efficacy in HI/HA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No study activity took place. The IND was withdrawn with the FDA by the Sponsor Investigator because of insurmountable hurdles in moving proposed research forward
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Lawson Wilkins Pediatric Endocrine Society (Other)
Responsible Party: Principal Investigator, Elizabeth A Rosenfeld, PI, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-018039
Record Dates: First submitted 2020-12-03; First posted 2021-08-02 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Hyperinsulinism-Hyperammonemia Syndrome
Keywords: hypoglycemia; hyperinsulinism; vitamin E
MeSH Terms: conditions — Hyperinsulinemic hypoglycemia, familial, 6; Hypoglycemia; Hyperinsulinism | interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Intervention Model Description: This single-group open-label dose-finding clinical study will use a before-and-after design, with repeated outpatient evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin E Dose-Escalation (Experimental): Subjects will take an oral Vitamin E (dl-alpha-tocopherol) supplement twice daily with a fat-containing meal for 6-9 weeks. The dose will be increased every 2-3 weeks over the course of the study (initial dose 600 IU twice daily, next dose 1,200 IU twice daily, final dose 2,400 IU twice daily). Formulations include softgel capsules in 200, 400, and 1,000 IU doses.
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Vitamin E — Twice daily oral supplementation with Vitamin E for 6-9 weeks.
  Other Names: dl-alpha-tocopherol

SUMMARY:
Congenital hyperinsulinism (HI) is a rare disorder of pancreatic beta cell insulin secretion that causes persistent and severe hypoglycemia starting at birth. Hyperinsulinism/hyperammonemia (HI/HA) syndrome is the second most common type of congenital HI and is caused by activating mutations in glutamate dehydrogenase (GDH). Patients with HI/HA exhibit fasting hyperinsulinemic hypoglycemia, protein-induced hypoglycemia, hyperammonemia, seizures, and intellectual disability independent of hypoglycemia. These effects result from abnormal GDH activity in the beta cells, liver and kidney cells, neurons, and astrocytes. The only available treatment for HI/HA syndrome is diazoxide, which acts on the beta cells to decrease insulin secretion but has no effect on GDH activity itself or on other cell types. Thus, there remains a significant unmet need for improved therapies for this disorder. Pre-clinical data show that vitamin E inhibits GDH activity in human cell lines and improves fasting hypoglycemia in a GDH HI mouse model. Pilot study data show that vitamin E supplementation with a moderate dose is well-tolerated in children and adults with HI/HA syndrome, while continuing diazoxide treatment. However, most subjects continued to exhibit protein-induced hyperinsulinemic hypoglycemia. We hypothesize that a higher vitamin E dose will inhibit GDH over-activity in subjects with HI/HA syndrome, resulting in improved hyperinsulinemic hypoglycemia, reduced blood ammonia concentration, and decreased seizure activity.

DETAILED DESCRIPTION:
The primary objective of this study is to determine an effective dose of vitamin E to reduce protein-induced hyperinsulinemia in subjects with HI/HA syndrome. Secondary objectives are to assess the effects of vitamin E on plasma C-peptide concentrations, serum alpha-tocopherol concentrations, blood ammonia concentrations, hypoglycemic events, and seizure frequency. The effect of vitamin E on brain glutamate levels and electroencephalogram findings will be explored.

This single-group open-label dose-finding clinical study will use a before-and-after design to compare clinical and laboratory data before and after 2-3 weeks of escalating doses of oral vitamin E treatment in subjects with HI/HA syndrome.

This single-site outpatient study will recruit up to 5 adult participants (18 years of age or older) with HI/HA syndrome.

Each study visit will consist of blood tests, an IV leucine acute insulin response (AIR) test, home glucose meter and continuous glucose monitor (CGM) review, and a symptom questionnaire. The baseline and final visits will also include electroencephalogram (EEG) and brain magnetic resonance imaging (MRI) with glutamate chemical exchange saturation transfer (GluCEST) analysis. After baseline assessments, including a 2 week run-in period of CGM use, subjects will take twice daily oral vitamin E (alpha-tocopherol) at home. After steady-state of that dose of vitamin E has been achieved (i.e. at least 2 weeks on the dose of vitamin E), subjects will return for the next study visit. If there is no dose-limiting toxicity, then the twice daily vitamin E dose will be increased, and the subjects will return for a subsequent study visit after at least 2 weeks. If there is no dose-limiting toxicity at this visit, then the twice daily vitamin E dose will be increased again, and the subjects will return for a final study visit after at least 2 weeks. If toxicity is identified at any point, vitamin E will be discontinued and final study visit procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥18 years.
* Diagnosis of HI/HA syndrome (based on glutamate dehydrogenase 1 [GLUD1] genetic test result and/or history of diazoxide-responsive hyperinsulinism with persistently elevated blood ammonia concentrations).
* Able to swallow softgels.
* Informed consent.

Exclusion Criteria:

* Vitamin E supplementation within 30 days prior to enrollment, including multivitamins containing vitamin E.
* Individuals who have experienced an allergic reaction to vitamin E.
* On concurrent therapy with a medication known to adversely interact with vitamin E.
* On concurrent therapy with a medication, supplement, or herbal remedy known to increase bleeding risk, including antiplatelet or anticoagulation therapy.
* Known increased risk of bleeding (coagulopathy, hemophilia, platelet defect, or platelet disorder) based on history, known or suspected vitamin K deficiency, baseline international normalized ratio (INR) >1.5, baseline prothrombin time (PT) >1.5 times the upper limit of normal, baseline partial thromboplastin time (PTT) >1.5 times the upper limit of normal, or baseline abnormal platelet function test result (VerifyNow-Aspirin <550 aspirin reactivity units [ARU], VerifyNow-adenosine diphosphate [ADP]/PRU <180 P2Y12 reaction units [PRU]).
* Known clotting disorder, including prior episodes of deep vein thrombosis or pulmonary embolism within the past 6 months.
* Evidence of severe hematologic abnormality including severe anemia (Hgb <10 g/dL) and/or thrombocytopenia (platelet count <150,000/mm3).
* Abnormal score on International Society on Thrombosis and Haemostasis (ISTH)-Bleeding Assessment Tool (>4 if male; >5 if female).
* Planned elective surgical procedure during study period.
* Evidence of a medical condition that might alter results or compromise the interpretation of results, including active infection, kidney failure, severe liver dysfunction, severe respiratory or cardiac failure.
* Any investigational drug use within 30 days prior to enrollment.
* Current use of somatostatin analog.
* Current adherence to a ketogenic diet.
* Pregnant or lactating females. Females must have a negative urine pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study and a minimum of 2 weeks after the last dose of study drug.
* Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Unable to provide informed consent (e.g. impaired cognition or judgment).
* Limited English proficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
protein-induced hyperinsulinemia | 4-11 weeks
  Change in plasma insulin concentration area under the curve (AUC) during leucine AIR test after vitamin E treatment compared to before.

SECONDARY OUTCOMES:
mean glucose concentration | 4-11 weeks
  Change in mean glucose concentration detected on continuous glucose monitor (CGM) during the study interval after vitamin E treatment compared to before.
proportion of time spent with glucose <70 mg/dL | 4-11 weeks
  Change in proportion of time spent with glucose <70 mg/dL, detected on continuous glucose monitor (CGM) during the study interval after vitamin E treatment compared to before.
proportion of time spent with glucose <50 mg/dL | 4-11 weeks
  Change in proportion of time spent with glucose <50 mg/dL, detected on continuous glucose monitor (CGM) during the study interval after vitamin E treatment compared to before.
hypoglycemic episodes | 4-11 weeks
  Change in frequency of hypoglycemic episodes (plasma glucose <70 mg/dL and plasma glucose <50 mg/dL) detected on home glucose meter and/or continuous glucose monitor (CGM) after vitamin E treatment compared to before.
protein-induced C-peptide release | 4-11 weeks
  Change in plasma C-peptide concentration area under the curve (AUC) during leucine AIR test after vitamin E treatment compared to before.
vitamin E | 4-11 weeks
  Change in serum alpha-tocopherol concentration after vitamin E treatment compared to before.
ammonia | 4-11 weeks
  Change in blood ammonia concentration after vitamin E treatment compared to before.
seizures | 4-11 weeks
  Change in frequency of seizures, based on symptom questionnaire, after vitamin E treatment compared to before.

OTHER OUTCOMES:
number of participants with EEG abnormalities | 8-11 weeks
  Change in brain electrical activity after vitamin E treatment compared to before.
brain glutamate | 8-11 weeks
  Change in glutamate concentration, as measured by brain GluCEST percent contrast, after vitamin E treatment compared to before.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Rosenfeld, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palladino AA, Stanley CA. The hyperinsulinism/hyperammonemia syndrome. Rev Endocr Metab Disord. 2010 Sep;11(3):171-8. doi: 10.1007/s11154-010-9146-0. PMID 20936362
- [Background] Snider KE, Becker S, Boyajian L, Shyng SL, MacMullen C, Hughes N, Ganapathy K, Bhatti T, Stanley CA, Ganguly A. Genotype and phenotype correlations in 417 children with congenital hyperinsulinism. J Clin Endocrinol Metab. 2013 Feb;98(2):E355-63. doi: 10.1210/jc.2012-2169. Epub 2012 Dec 28. PMID 23275527
- [Background] Hsu BY, Kelly A, Thornton PS, Greenberg CR, Dilling LA, Stanley CA. Protein-sensitive and fasting hypoglycemia in children with the hyperinsulinism/hyperammonemia syndrome. J Pediatr. 2001 Mar;138(3):383-9. doi: 10.1067/mpd.2001.111818. PMID 11241047
- [Background] Kelly A, Ng D, Ferry RJ Jr, Grimberg A, Koo-McCoy S, Thornton PS, Stanley CA. Acute insulin responses to leucine in children with the hyperinsulinism/hyperammonemia syndrome. J Clin Endocrinol Metab. 2001 Aug;86(8):3724-8. doi: 10.1210/jcem.86.8.7755. PMID 11502802
- [Background] Stanley CA, Baker L. Hyperinsulinism in infancy: diagnosis by demonstration of abnormal response to fasting hypoglycemia. Pediatrics. 1976 May;57(5):702-11. PMID 940710
- [Background] Li M, Smith CJ, Walker MT, Smith TJ. Novel inhibitors complexed with glutamate dehydrogenase: allosteric regulation by control of protein dynamics. J Biol Chem. 2009 Aug 21;284(34):22988-3000. doi: 10.1074/jbc.M109.020222. Epub 2009 Jun 15. PMID 19531491
- [Background] Treberg JR, Clow KA, Greene KA, Brosnan ME, Brosnan JT. Systemic activation of glutamate dehydrogenase increases renal ammoniagenesis: implications for the hyperinsulinism/hyperammonemia syndrome. Am J Physiol Endocrinol Metab. 2010 Jun;298(6):E1219-25. doi: 10.1152/ajpendo.00028.2010. Epub 2010 Mar 23. PMID 20332361
- [Background] Ferslew KE, Acuff RV, Daigneault EA, Woolley TW, Stanton PE Jr. Pharmacokinetics and bioavailability of the RRR and all racemic stereoisomers of alpha-tocopherol in humans after single oral administration. J Clin Pharmacol. 1993 Jan;33(1):84-8. doi: 10.1002/j.1552-4604.1993.tb03909.x. PMID 8429120